CLINICAL TRIAL: NCT05189626
Title: Effectiveness of Kaltenborn Mobilizations Versus Muscle Energy Technique in Adhesive Capsulitis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Health Education Research Foundation (HERF) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 142/IREF/RMU/2021
Record Dates: First submitted 2021-12-11; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Adhesive Capsulitis of Shoulder
Keywords: Adhesive Capsulitis,Mobilizations, muscle energy technique
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: There are two groups Group 1 and 2.Group 1 is treated with Muscle energy techniques and Group 2 is treated with kaltenborn mobilizations for 30 minutes per session,3 days per week for 4 weeks.
Who Masked: Participant, Care Provider
Masking Description: It is a single blinded study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Muscle energy technique
  Interventions: Other: Muscle energy technique
- Group B (Experimental): Kaltonborn mobilizations
  Interventions: Other: Kaltonborn mobilizations

INTERVENTIONS:
Other: Muscle energy technique — Post Isometric relaxation(muscle energy technique) 3 days/ week for 4 weeks
  Arms: Group A
Other: Kaltonborn mobilizations — Kaltonborn mobilizations grade II and III will be performed on Glenohumeral joints 3 days/ week for 4 weeks.
  Arms: Group B

SUMMARY:
Total of 30 patients are selected according to inclusion criteria by convenient sampling and randomly allocated by sealed envelop method into two groups. Group 1 is treated with Muscle energy technique(Post isometric relaxation) and Group 2 is treated with Grade II,III Kaltenborn mobilizations and both groups also receives conventional therapy in form of Codman exercise and Wall ladder exercises.Data will be collected at baseline then after 2 weeks and after 4 weeks of intervention.

DETAILED DESCRIPTION:
The purpose of study is to determine effectiveness of muscle energy techniques(Post Isometric relaxation) and Kaltenborn mobilizations and to compare the effectiveness of both techniques on pain and functional disability in patients with Adhesive capsulitis.Several studies about the effects of Maitland mobilizations and Muscle energy technique have been conducted. Evidence regarding the comparison of Kaltenborn mobilizatuons and post isometric relaxation is sparse. There has been no work regarding effectiveness of these two techniques in improving pain and functional disability in patients of Adhesive capsulitis.

Kaltonborn Mobilizations involves the application of a passive sustained stretch technique to enhance joint mobility without articular surface suppression. The forces applied to increase joint mobility are graded from I-III. Grade I applies a distraction of minor intensity that hardly causes stress within the joint capsule; it is often used to decrease pain. Grade II refers to a force that stretches the periarticular tissue; such stimulus is colloquially referred to as "taking up the slack." Finally, Grade III force causes enough distraction or gliding so that joint capsule can sufficiently stretch; it is often used for enhancing ROM.

MET is unique in its application as the client provides the initial effort while the practitioner facilitates the process. One of the main uses of this method is to normalize joint range, rather than increase flexibility, and techniques can be used on any joints with restricted Range of Motion (ROM) identified during the passive assessment. The main effects of MET can be explained by two distinct physiological processes: Post Isometric Relaxation (PIR) and Reciprocal Inhibition (RI). Post isometric contraction decrease muscle tone in single group of muscle after brief period of submaximal isometric contraction of same muscle.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 60 years.
* Duration of complaint for more than 3 months.
* Gender: Both Male and Female.
* Patients with idiopathic frozen shoulder
* Patients having restriction in more than 2 ranges
* Patients with diabetes

Exclusion Criteria:

* Shoulder dislocation, fracture or labral tear.
* Shoulder girdle motor control deficit associated with neurological disorder.
* Any bony deformities acquired or congenital in glenohumeral joint.
* Patients with language barrier.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Shoulder pain and disability index | 4 weeks
  Shoulder pain and disability index is used to measure pain and functional disability level. Total scores range from 0 to 130 with a percentage score of 0 indicating less shoulder disability and 100 indicating more shoulder dysfunction
Universal goniometer | 4 weeks
  universal goniometer is used to measure shoulder range of motion.

CONTACTS AND LOCATIONS:
Overall Officials: Aqsa Anwar, DPT, Principal Investigator — Rawalpindi Medical College
Locations (1):
- Holy family hospital, Rawalpindi, Punjab Province, Pakistan